CLINICAL TRIAL: NCT03708731
Title: Exploring Adherence Monitoring in Sickle Cell Disease
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ExAMS
Record Dates: First submitted 2018-10-04; First posted 2018-10-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Youth; Hydroxyurea; Non-Adherence; Electronic Adherence Monitoring; AdhereTech smart bottle
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle Cell Disease: All participants who meet eligibility requirements and consent to the study.

SUMMARY:
Despite the well-documented benefits of hydroxyurea (HU) therapy in decreasing morbidity and mortality in youth with Sickle cell disease (SCD), pediatric HU adherence rates range as low as 49% and lead to discontinuation of HU regimens in 8-20%. In addition, treatment non-adherence may lead to unnecessary increases in medication dosage resulting from erroneous assumption that a patient is non-responsive to treatment (versus non-adherent to the regimen as prescribed). Given the detrimental effects of non-adherence, assessment of and intervention for HU non-adherence is essential to improving health outcomes in the pediatric SCD population.

Electronic adherence monitoring is widely considered the "gold standard" in objective adherence measurement. These monitors provide continuous, real- time records of medication adherence and reveal problematic behavior patterns, including underdosing, overdosing, delayed dosing, "drug holidays," and "white coat" adherence. Overall, electronic adherence measures are considered valid, reliable, and accurate, with clear advantages over pharmacy refill records, physician estimates and self-report measures.

The primary purpose of this pilot study is to determine the use of the AdhereTech as a feasible and valid measure of HU adherence in pediatric SCD.

Primary Objective Estimate the association between HU adherence as measured by the AdhereTech device to a) caregiver-report, b) youth-report, c) lab values, d) pill- count, and e) Medication Possession Ratio (MPR) adherence measures Secondary Objectives Estimate the rate of consent to the study, the rate of AdhereTech device use, the rate of AdhereTech device failure, and the perceived acceptability of using the AdhereTech device, as reported by caregivers and youth

DETAILED DESCRIPTION:
The AdhereTech smart bottle is an electronic medicine dispenser with a tracking and reminder system connected wirelessly. The device provides real time adherence aids to the patient and this information is relayed to the provider. The device can sense the amount of pills remaining inside the bottle. This information is measured periodically and concurrently sent to a secure database using cellular data technology. Thus, AdhereTech bottles can be used to determine whether medication was removed from the bottle, the amount of medication removed, and the timing of removal.

Participants ages 12.0-17.99 who are receiving HU prescribed in pill form will use the AdhereTech smart bottle for a two-month period. Participants and their caregivers will complete self-report measures of adherence at the baseline, 1 month and 2 month clinic visits, a Demographic questionnaire at the baseline clinic visit and an Acceptability questionnaire at the 1 month and 2 month clinic visits using Audio Computer-Assisted Self-Interviews (ACASI) on a password protected laptop.

Lab values and clinical information will be obtained through medical records review and adherence information from pill counts and pharmacy records.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCD (any genotype)
* Ages 12.0 - 17.99 at time of study enrollment
* Stable HU dose composed of only one capsule strength prescribed in pill formulation for ≥ 6 months without documented hematological toxicity (excluding dose adjustments for weight gain)
* Lives with their legal guardian
* Anticipated to return to clinic at proposed 4-week intervals

Exclusion Criteria:

* Primary caregiver and/or youth unable to understand English and/or youth not cognitively intact (known IQ < 70) such that the study questionnaire cannot be understood and completed.
* Participant unable to complete the questionnaires due to refusal or current acute illness (e.g., pain crisis).
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants ages 12.0-17.99 with Sickle cell disease any genotype and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the association between AdhereTech device HU adherence to caregiver-report of adherence | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). Caregiver-report of their child's HU adherence will be assessed by the Medical Adherence Measure (MAM), a measure of 7-day self-reported adherence. Each subject's caregiver-reported adherence will be calculated as: [(medication reported taken [(medication reported taken ÷ medication prescribed) x 100]. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with the caregiver-report of their child's adherence.
Estimate the association between AdhereTech device HU adherence to youth-reported adherence | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). Youth-report of their HU adherence will be assessed by the Medical Adherence Measure (MAM), a measure of 7-day self-reported adherence. Each subject's self-reported adherence will be calculated as: [(medication reported taken [(medication reported taken ÷ medication prescribed) x 100]. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with the youth-reported adherence.
Estimate the association between AdhereTech device HU adherence to fetal hemoglobin (HbF) lab values | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). We will extract fetal hemoglobin (HbF; g/dl) lab value from each subject's medical record. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with the fetal hemoglobin (HbF) lab value.
Estimate the association between AdhereTech device HU adherence to mean corpuscular volume (MCV) lab values | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). We will extract mean corpuscular volume (MCV; L) lab value from each subject's medical record. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with the mean corpuscular volume (MCV) lab value .
Estimate the association between AdhereTech device HU adherence to the Medication Possession Ratio (MPR) | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). Medication Possession Ratio (MPR) will be calculated as: [(number of days medication in family's possession ÷ number of days for which medication prescribed) x 100]. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with the Medication Possession Ratio (MPR).
Estimate the association between AdhereTech device HU adherence to pill count | Continuous over two months, baseline to off study
  For each subject, we will calculate the proportion of days of opening the AdhereTech device across the two month study period (days with missing information will not be counted). We will calculate each subject's pill count adherence as: [(number of pills removed ÷ medication prescribed) x 100]. We will estimate the Spearman's rank-based correlation, with 95% confidence interval, of the AdhereTech device adherence with pill count adherence.

SECONDARY OUTCOMES:
Estimate rate of consent to the study | Once, at baseline
  We will descriptively examine rate of refusal and study participation: (Number participants consented ÷ Total families approached) x 100%
Estimate rate of AdhereTech device use | Continuous over two months, baseline to off study
  We will descriptively examine rate of AdhereTech device use: (Number participants keeping medication in device during entire trial ÷ Total participants) x 100%
Estimate rate of AdhereTech device failure | Continuous over two months, baseline to off study
  We will descriptively examine AdhereTech device failure (i.e., a device does not register openings as verified by study staff at the time device is returned to study team): (Number devices failing ÷ Total devices) x 100%
Estimate the perceived acceptability of using the AdhereTech device, as reported by caregivers and youth | Continuous over two months, baseline to off study
  We will descriptively examine reported acceptability of using the AdhereTech device: Point estimation and interval estimations for the counts and frequencies of favorable responses of acceptability will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jerlym Porter, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols